CLINICAL TRIAL: NCT05412667
Title: Investigation of TWK10 Administration on the Effects of Amino Acid Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chi-Chang Huang (Other)
Collaborators: Synbio Tech Inc. (Industry)
Responsible Party: Sponsor-Investigator, Chi-Chang Huang, PI, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 21-035-B1
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Amino Acid; Exercise; Probiotic; Body Composition
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Pea protein without TWK10 (20g/day)
  Interventions: Other: Placebo
- TWK10 (Experimental): Pea protein (20g/day) with TWK10 (10 billion CFU/day)
  Interventions: Dietary Supplement: TWK10

INTERVENTIONS:
Dietary Supplement: TWK10 — 1. 4 days without training: drink 2 hours before bedtime.
  2. 3 days of training: drink within 30 minutes after training (uniformly brewed in the laboratory).
  3. To analyze the amino acid concentration in blood, drink it immediately before blood collection.
  Arms: TWK10
Other: Placebo — 1. 4 days without training: drink 2 hours before bedtime.
  2. 3 days of training: drink within 30 minutes after training (uniformly brewed in the laboratory).
  3. To analyze the amino acid concentration in blood, drink it immediately before blood collection.
  Arms: Placebo

SUMMARY:
The most common problem among sports people is that no matter how much protein food or products they eat, their sports performance cannot be improved, resulting in failure to achieve breakthroughs in sports performance. The cause of the trouble is digestion and absorption problems. The key is intestinal problems. If gastrointestinal function is maintained in a healthy state, then exercise performance must be maintained at a considerable level. Therefore, how to choose the source of protein in the diet is one of the most concerned issues of the sports crowd. Although past studies have confirmed that the essential amino acids in animal protein can be absorbed and utilized better than plant protein, plant protein can be broken down into easily digestible peptides and amino acids by pepsin. Promote the metabolite pool in the large intestine and the amino acid balance of the host in the small intestine. Recent studies have pointed out that the proteases and peptidases in lactic acid bacteria can provide free amino acids for the best growth of bacteria, and can increase the distribution of amino acids in the blood, the speed of muscle synthesis and the content of branched chain amino acids. However, the mechanism of action of Lactobacillus plantarum on protein digestion and amino acid absorption in the host is still unclear. Therefore, the purpose of this study is to explore the effect of supplementing sports lactic acid bacteria TWK10 in human experiments to effectively improve the amino acid bioabsorption rate of plant protein supplements. 40 subjects were randomly divided into 2 groups, each with 20 people (male and female): (1) pea protein without TWK10 (placebo), (2) TWK10 group (TWK10). The two groups of subjects were supplemented with test samples for 28 consecutive days and performed paired sports training 3 times a week. Before and after the intervention, the samples were subjected to exercise testing, blood and fecal sample collection, body composition analysis, and muscle mass analysis.

ELIGIBILITY:
Inclusion Criteria:

* Have exercise habits (exercise at least 3 times a week for at least 30 minutes each time),
* Healthy body

Exclusion Criteria:

* Smoking
* Alcohol consumption
* Cardiovascular disease
* Neuromuscular disease
* Metabolic disease
* Asthma, pregnant or breastfeeding
* BMI>27
* Allergic to peanuts .

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Amino acid | From Baseline to 4 Weeks Assessed, including time point: baseline, 30 minutes, 60 minutes, 120 minutes, and 180 minutes post ingestion)
  Liquid chromatography tandem mass spectrometry (LC-MS/MS) was used for analysis, wherein the liquid chromatography system was Acquity UPLC, and the column used was Waters C18 column (2.1 × 150 mm, 1.8 μm), and the temperature of the column was set at 45 °C, the mobile phases used were water and 100% acetonitrile, both of which contained 0.1% formic acid, the flow rate was 0.6 mL/min, and the injection volume of the test solution was 2 μL.
Muscle composition | From Baseline to 4 Weeks Assessed
  Use muscular ultrasound (BenQ T3300) to scan
Isometric Mid-Thigh Pull (IMTP) | From Baseline to 4 Weeks Assessed
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak force (PF) were recorded.
Isometric Mid-Thigh Pull (IMTP) | From Baseline to 4 Weeks Assessed
  Customized IMTP test equipment and two force plates (type 9287BA, Kistler Instruments AG, Winterthur, Switzerland) were used. All participants stood with their feet the same width apart, and the rod was placed between the thighs, with the torso upright, the spine neutral, and the knee and hip angles at 140°, to familiarize the participants with the IMPT test method. The average absolute peak rate of force development (RFD) parameters were recorded.
Wingate Anaerobic Test (WAnT) | From Baseline to 4 Weeks Assessed
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The recorded results were the relative mean power (W/kg)
Wingate Anaerobic Test (WAnT) | From Baseline to 4 Weeks Assessed
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The recorded results were the relative peak power (W/kg)
Wingate Anaerobic Test (WAnT) | From Baseline to 4 Weeks Assessed
  After a standard warm-up, all subjects were assessed with the classical WAnT on a cycloergometer (Monark 894E, Varberg, Sweden) in a 30 s "go all out" ultramax test. The seat height was adjusted to the satisfaction of each participant, and toe clips prevented the feet from slipping off the pedals. Before the initial test, the subjects warmed up for 5 min, and the power was approximately 50 W. After the warm-up, two preparation exercises lasting 3 s, during which the actual test load was 3% of their own body weight, were applied to accustom the participant to resistance. The test started, and the resistance was set on the friction belt of the dynamometer. External loading was estimated individually at 5% body weight. The recorded results were the fatigue index (%)
dual-energy X-ray absorptiometry, DXA | From Baseline to 4 Weeks Assessed
  A non-invasive dual-energy X-ray absorptive bone density testing room (Lunar iDXA, GE Healthcare, Chicago, IL, USA) was used for systemic body composition and bone density measurements. The subject was required to lie flat on the test bed, with their body at the center line, and their limbs within the detection range. Two different energy X-rays were used to scan the inspected part, then the scintillation detector received the X-rays that had penetrated the inspected part, and analyzed the obtained muscle mass
dual-energy X-ray absorptiometry, DXA | From Baseline to 4 Weeks Assessed
  A non-invasive dual-energy X-ray absorptive bone density testing room (Lunar iDXA, GE Healthcare, Chicago, IL, USA) was used for systemic body composition and bone density measurements. The subject was required to lie flat on the test bed, with their body at the center line, and their limbs within the detection range. Two different energy X-rays were used to scan the inspected part, then the scintillation detector received the X-rays that had penetrated the inspected part, and analyzed the obtained fat mass
Bench press test | From Baseline to 4 Weeks Assessed
  Bench press with Smith machine and add weight to find individual 1RM

SECONDARY OUTCOMES:
Checklist Individual Strength (CIS) questionnaire | From Baseline to 4 Weeks Assessed
  Assessing subjects' living conditions using the CIS scale. 1 is the least match, 5 is the most match
Visual Analog Fatigue Scale (VAFS) | From Baseline to 4 Weeks Assessed
  Using the VAS scale to measure the subjective feelings of the subjects after exercise, 1 is the least tired, 5 is the most tired
Rating of Perceived Exertion (RPE) scale | From Baseline to 4 Weeks Assessed
  Use the RPE scale to record how hard the subjects are after the test, 6 points are the least hard, 20 points are the hardest
3-day dietary recording four weeks | From Baseline to 4 Weeks Assessed
  After 4 weeks of intervention, the 3-day diet was recorded and the calorie intake was calculated by the dietitian

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Institute of Sports Science, National Taiwan Sport University, Taoyuan District, Taiwan